CLINICAL TRIAL: NCT04680377
Title: Using Microbiome to Predict Durvalumab Toxicity in Post-CCRT NSCLC Patients (Microdurva)
Brief Title: Using Microbiome to Predict Durvalumab Toxicity in Post- Concurrent Chemoradiation Therapy (CCRT) NSCLC Patients
Acronym: Microdurva
Status: Recruiting | Type: Observational
Sponsor: Jun Zhang, MD, PhD (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, MD, PhD, MD, PhD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: IIT-2019-AZmicrobiome
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: NSCLC, Stage III; Locally Advanced Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal and buccal swabs, and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving standard of care durvalumab: Prior to receiving treatment participants will have samples taken from three different sources to test the microbiome bacteria to determine if it will help predict toxicity to the treatment

SUMMARY:
This phase IV study is hoping to determine if examining the microbiome in non-small cell lung cancer participants who will receive durvalumab can predict treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Life expectancy ≥12 weeks
* Males and females age ≥ 18 years
* Allowable type and amount of prior therapy:

Participants must have received two or more cycles of platinum-based chemotherapy (containing etoposide, vinblastine, vinorelbine, a taxane [paclitaxel or docetaxel], or pemetrexed) concurrently with definitive radiation therapy (54-66 Gy)

* Eastern Cooperative Oncology Group (ECOG) Performance Status = 0 or 1
* Body weight >30 kg (66.14 lbs)
* Participants must have histologically- or cytologically-documented NSCLC who present with locally advanced, unresectable (Stage III) disease
* Participants must have not progressed following definitive, platinum-based, concurrent chemoradiation therapy
* Adequate organ function based on laboratory results
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use an acceptable form of contraception for the duration of study participation, and for the time specified following completion of therapy

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or if the participant is in the follow-up period of an interventional study
* Participation in another clinical study with an investigational product during the last 4 weeks prior to enrollment on this study
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment
* Mixed small cell and non-small cell lung cancer histology
* Participants who receive sequential chemoradiation therapy for locally advanced NSCLC
* Participants with locally advanced NSCLC who have progressed whilst definitive platinum based, concurrent chemoradiation therapy
* Receipt of any investigational drug within 4 weeks prior to the first dose of durvalumab; and in the case of monoclonal antibodies (not immunotherapy) 6 weeks prior to the first dose of durvalumab
* Participants who have received prior anti-programmed death (PD)-1, anti- programmed death ligand (PD-L)1 or anti- cytotoxic T-lymphocyte-associated protein (CTLA)-4
* Participants who have received prior immunotherapy
* Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product (IP). Note: Participants, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of IP
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab
* Any unresolved toxicity CTCAE ≥ Grade 2 from the prior chemoradiation / anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Any grade pneumonitis from prior chemoradiation therapy
* Active infection
* Recent major surgery within 28 days prior to the first dose of study therapy
* Active or prior documented autoimmune or inflammatory disorders
* History of primary immunodeficiency
* History of another primary malignancy
* History of allogenic organ transplantation/organ transplant that requires therapeutic immunosuppression
* History of leptomeningeal carcinomatosis
* Participants with active ventricular arrhythmia requiring medication
* Uncontrolled intercurrent illness
* Participants who have progressed following definitive, platinum-based, concurrent chemoradiation therapy
* Known allergy or hypersensitivity to durvalumab or any of durvalumab's excipients
* Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have histologically- or cytologically-documented NSCLC who present with locally advanced, unresectable (Stage III) disease.
  Participants must have not progressed following definitive, platinum-based, concurrent chemoradiation therapy.
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or higher adverse events (AE's) | Up to 18 months
  CTCAE 5.0
Longitudinal changes in Microbiome | Up to 18 months from study start
  Metagenomic sequencing and taxonomic analysis
Longitudinal changes in bacterial metabolic pathway | Up to 18 months from study start
  Metagenomic sequencing and Kyoto Encyclopedia of Genes and Genomes (KEGG) mapping

SECONDARY OUTCOMES:
Time-to-treatment withheld due to AEs | Up to 18 months from study start
  Time measured by days
Time to immune-mediated AEs requiring systemic intervention | Up to 18 months from study start
  Time measured by days
Progression free survival | Up to 36 months from study start
  Time measured by months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Principal Investigator — The University of Kansas Cancer Center
Locations (2):
- United States (2):
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - Rhode Island Hospital, Brown University, Providence, Rhode Island

REFERENCES:
- [Background] Swami U, Zakharia Y, Zhang J. Understanding Microbiome Effect on Immune Checkpoint Inhibition in Lung Cancer: Placing the Puzzle Pieces Together. J Immunother. 2018 Oct;41(8):359-360. doi: 10.1097/CJI.0000000000000232. PMID 29781826
- [Background] Strouse C, Mangalam A, Zhang J. Bugs in the system: bringing the human microbiome to bear in cancer immunotherapy. Gut Microbes. 2019;10(2):109-112. doi: 10.1080/19490976.2018.1511665. Epub 2018 Sep 5. PMID 30183502